CLINICAL TRIAL: NCT06027099
Title: Integrating Tailored Postoperative Opioid Tapering and Pain Management Support for Patients on Long-Term Opioid Use Presenting for Spine Surgery
Brief Title: CARES-Spine (Comprehensive Analgesic, Recovery, and Education Support for Spine Surgery) Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71909
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Back Pain; Neck Pain; Opioid Misuse
MeSH Terms: conditions — Chronic Pain; Back Pain; Neck Pain; Opioid-Related Disorders | interventions — tizanidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MI-Opioid Taper and tizanidine (Experimental)
  Interventions: Drug: Tizanidine; Behavioral: MI-Opioid Taper
- MI-Opioid Taper and placebo (Experimental)
  Interventions: Behavioral: MI-Opioid Taper; Drug: Placebo
- Enhanced Usual Care (Active Comparator)
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Drug: Tizanidine — Tizanidine 2mg three times a day for 5 weeks after surgery
  Arms: MI-Opioid Taper and tizanidine
Behavioral: MI-Opioid Taper — Motivational Interviewing (MI) and guided Opioid Tapering support adapting MI principles for enhancing motivation to change in pain treatment and tailoring key MI tools to postoperative opioid use delivered through weekly phone calls from weeks 2 to 7, and at week 11. The guided opioid tapering protocol will be a 25% total daily opioid dose reduction every 7 days with opioid discontinuation 7 days after reaching 1 opioid pill per day.
  Arms: MI-Opioid Taper and placebo; MI-Opioid Taper and tizanidine
Drug: Placebo — 1 tablet three times a day for 5 weeks after surgery
  Arms: MI-Opioid Taper and placebo
Behavioral: Enhanced Usual Care — Participants will receive weekly phone calls from weeks 2 to 7, and at week 11. 1 topic per call will be reviewed in this sequence:1) standardized instructions on taking opioid medications after surgery, 2) safe opioid use, 3) avoiding medication errors, 4) local mental health resources and 988 Suicide & Crisis lifeline, 5) disposal of unused medications, 6) prescription drug abuse, and 7) complementary health approaches for chronic pain. Education materials will be reviewed in a didactic style without a tailored discussion.
  Arms: Enhanced Usual Care

SUMMARY:
Three-arm randomized controlled trial, of Motivational Interviewing and guided Opioid Tapering support (MI-Opioid Taper) and tizanidine vs. MI-Opioid Taper and placebo vs. enhanced usual care to promote postoperative opioid cessation and pain cessation and reduce the incidence of postoperative opioid misuse among patients undergoing spine surgery.

DETAILED DESCRIPTION:
In this Type 1 hybrid effectiveness-implementation three-arm parallel RCT, 375 patients with preoperative LTOU undergoing spine surgery will be recruited across 4 sites (Stanford, Harvard, Wake Forest, U. of Kansas) and randomized to 1 of 3 groups (MI-Opioid Taper and tizanidine, MI-Opioid Taper and placebo, enhanced usual care) and followed for 12 months. The primary outcome is time to baseline opioid use. Secondary outcomes are time to opioid cessation, opioid dispensing cessation, pain cessation, and risk of postoperative opioid misuse. We will examine motivation for change, change talk, and reduction in pain as mediators of treatment effects and characterize treatment interactions with participant attributes in predicting both treatment engagement and efficacy. A mixed-methods evaluation using the RE-AIM framework will explore barriers and facilitators to future larger-scale implementation of MI-Opioid Taper. The project will address the unmet needs of patients on long-term opioid use presenting for surgery in need of precision postoperative pain care to minimize opioid-related harms.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-64 scheduled for elective spine surgery for lumbar or cervical degenerative disease (e.g. lumbar or cervical disc herniation, lumbar or cervical spinal stenosis, lumbar or cervical degenerative spondylolisthesis, lumbar or cervical disc degeneration, or degenerative cervical myelopathy including cervical spondylotic myelopathy).

  * Preoperative long-term opioid use (Defined as ≥ 90-day duration of use in the 4 months preceding surgery either via self-report or state PDMP.
  * Participants must report at least one of the following on preoperative assessments:

Current Opioid Misuse Measure (COMM) score greater than or equal to 9 Answering "Yes" to any of the following items on the modified Brief Pain Inventory (BPI)1) Over the past 24 hours have you needed to take your pain medication to help you sleep; 2)Have you taken any pain medications for any reason other than your pain, such as to reduce anxiety or improve mood? 3) Have you taken more pain medication than was prescribed to you in the past 24 hours? Score of greater than or equal to 2 on any Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) item Positive Alcohol Use Disorders Identification Test (AUDIT-C) score (greater than or equal to 4 for men, greater than or equal to 3 for women)

* Elevated opioid use 14 days after surgery compared to baseline daily OME Defined as average daily OME assessed over 3 days 1 week before surgery compared to average daily OME reported on postoperative days 12 to 14 to account for as-needed dosing and day-to-day variations in opioid use.
* English-speaking
* Ability and willingness to complete online assessments

Exclusion Criteria:

* Infection, tumor, or fracture at the operative site
* Allergy or intolerance to tizanidine
* Current use of tizanidine
* Renal impairment
* Hepatic impairment including cirrhosis or elevated enzymes
* Concurrent use of other α2-adrenergic agonists, skeletal muscle relaxants
* Concurrent use of: fluvoxamine, ciprofloxacin,zileuton, fluoroquinolones, antiarrhythmics (amiodarone, mexiletine, propafenone, verapamil), cimetidine, famotidine, oral contraceptive pills, acyclovir, ticlopidine, and fexinidazole
* Pre-existing hypotension, sedation, dizziness, severe respiratory insufficiency.
* Opioid Use Disorder
* Suicidality as assessed by the Patient Health Questionnaire-9 (PHQ-9) Question 9 score ≥ 1
* Pregnancy, breastfeeding, or planning to conceive
* Cancer diagnosis, active malignant neoplasm (metastatic or local) or evidence of paraneoplastic syndrome
* Conditions causing inability to complete assessments (education, cognitive ability, mental status, medical status)
* Participating in another clinical trial with an active treatment arm

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Time to baseline opioid use | Assessed after surgery up to 1 year after surgery
  Defined as the 1st of 2 consecutive reports of return to preoperative daily OME use or lower on the modified BPI.Preoperative daily OME use is defined as average daily OME assessed over 3 days, on days 7 to 9 before surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No